CLINICAL TRIAL: NCT01526395
Title: Decreasing the Use of Unmodified ECT in an Indian Hospital
Brief Title: Decreasing the Use of Unmodified Electroconvulsive Therapy (ECT) in an Indian Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); Chhatrapati Shahuji Maharaj Medical University (Other)
Responsible Party: Principal Investigator, Irving Reti, Associate Professor, Johns Hopkins University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NA_00027421
Record Dates: First submitted 2011-12-21; First posted 2012-02-03 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Schizophrenia
Keywords: electroconvulsive therapy; ECT; unmodified; anesthesia; propofol
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Schizophrenia | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unmodified ECT (No Intervention): Data will be collected on patients receiving ECT in its unmodified form prior to the introduction of low dose propofol sedation.
- Low Dose Propofol (Active Comparator): Subjects will be given low dose propofol prior to ECT.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — The major intervention proposed in this study is the introduction of low dose IV propofol for sedation prior to ECT treatment at C.S.M Medical University. The investigators will use a dose of 0.25 to 0.50 mg/kg of IV propofol. The maximum dose of 0.50 mg/kg is not sufficient for anesthesia (i.e., to make unconscious), but should provide a light level of sedation and be "amnestic," meaning the patient should have memory loss for the period of time around the ECT procedure itself. The propofol dose will be titrated upwards (from an initial dose of 0.25 mg/kg) with successive treatments in increments of 0.05mg/kg, until it is just sufficient to be lightly sedating. ECT will be administered 30 to 60 seconds after propofol is injected. ECT may be given up to three times per week.
  Arms: Low Dose Propofol

SUMMARY:
In developing countries, electroconvulsive therapy (ECT) is typically delivered without the use of an anesthetic prior to the treatment, known as unmodified ECT. This interventional study aims to decrease the practice of unmodified ECT at Chhatrapati Shahuji Maharaj Medical University, U.P. & G.M. & Associated Hospitals (C.S.M) by administering a low dose anesthetic (propofol) prior to ECT delivery. In so doing, the investigators hope to facilitate the transition from unmodified to modified ECT without incurring excessive costs to the center. It is hypothesized that ECT patients will opt for modified treatment, that adverse effects will be minimal, and that costs will not rise prohibitively.

DETAILED DESCRIPTION:
Patients that are currently receiving unmodified ECT at C.S.M Hospital will be eligible for the first phase of the study in which only data is collected. Three months after study start, patients who are to receive ECT for a psychiatric disorder will be eligible to participate in the intervention (introduction of propofol at a low dose prior to ECT). Data collection will include information such as demographics, ratings scales, seizure length, anxiety level, adverse events, and number of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are any psychiatric patients at C.S.M. for whom ECT is recommended by their doctor, whether or not they actually receive ECT.
* Subjects must also have an American Society for Anesthesiologists (ASA) rating score of 1 (completely healthy) or 2 (mild systemic disease) with stable symptoms and laboratory values.
* Subjects must be between the ages of 18 to 65 years old and be able to give informed consent.

Exclusion Criteria:

* Patients who speak neither English nor Hindi.
* History of or anatomical evidence for a difficult airway being a short mandible, micrognathia, large tongue or large goiter, arthritis of the jaw or neck, or enlarged tonsils. For this reason we will also exclude patients with a BMI > 28.
* Respiratory tract disease including asthma, respiratory infection, chest wall disease, chronic obstructive pulmonary disease, obstructive sleep apnea, or other disorder which might compromise the airway. Patients who smoke 15 or more cigarettes per day will be excluded unless abstinent for at least 10 days, to reduce the risk of respiratory complications.
* Patients who receive modified ECT during the first phase of the study.
* Pregnant women or women who are breastfeeding.
* Hypersensitivity to propofol or any of its components.
* Patients who are hemodynamically unstable or who have impaired cardiac function.
* BMI < 18.
* Patients with a history of epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients receiving ECT who agree to the modified form of treatment after it is offered. | 6 months

SECONDARY OUTCOMES:
Rate at which ECT is offered and refused. | 6 months
Change in patient anxiety measured by the state portion of the State-Trait Anxiety Inventory. | Baseline and completion of ECT treatments or up to 6 months, whichever comes first
Inpatient length of stay calculated from onset of ECT administration. | 6 months
Number of ECTs required to complete a course of treatment | 6 months
Changes in scales used to assess severity of symptoms. The investigators will record changes in the Hamilton Depression Rating Scale, the Young Mania Rating Scale, the Brief Psychiatric Rating Scale and the Clinical Global Impression Severity scale. | Baseline and completion of ECT treatments or up to 6 months, whichever comes first
Cognitive changes, monitored by the Mini Mental State Examination (MMSE) | Baseline and completion of ECT treatments or up to 6 months, whichever comes first
Monitoring of adverse effects such the occurence of emergent delirium, headaches, muscle aches, nausea and vomiting, and fractures and dislocations. | Baseline and completion of ECT treatments or up to 6 months, whichever comes first
Monitoring of delirium using the test with the Confusion Assessment Method for the ICU (CAM-ICU). | Baseline and completion of ECT treatments or up to 6 months, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Irving M Reti, MBBS, Principal Investigator — Johns Hopkins University
Locations (1):
- Chhatrapati Shahuji Maharaj Medical University, U.P. & G.M. & Associated Hospitals, Lucknow, Uttar Pradesh, India